CLINICAL TRIAL: NCT05762016
Title: A Comparison of the Outcomes of a Novel Technique of Mini- Incision and Self-Express (MISE) for Breast Abscess With the Conventional Techniques: A Retrospective Comparative Cohort Study
Brief Title: Outcomes of a Novel Technique of Mini- Incision and Self-Express (MISE) for Breast Abscess
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB Ref:2021/2634
Record Dates: First submitted 2023-02-22; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Breast Infection
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- incision and drainage group: patients with breast abscess who undergo incision and drainage
- percutaneous drainage group: patients with breast abscess who undergo percutaneous drainage
- MISE group: patients with breast abscess who undergo MISE
  Interventions: Procedure: Bedside Mini-Incision and Self-Express (MISE)

INTERVENTIONS:
Procedure: Bedside Mini-Incision and Self-Express (MISE) — To perform bedside mini incision and encourage patients to self express the pus following the intervention
  Groups: MISE group

SUMMARY:
Conventional techniques for treatment of breast abscess, such as incision and drainage/percutaneous drainage, have disadvantages. Bedside Mini-Incision and Self-Express (MISE) is a novel technique for breast abscess. The outcomes of MISE were compared to the conventional techniques.

DETAILED DESCRIPTION:
outcomes such as recovery time, duration of antibiotics use etc will be compared between the various groups of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathologically confirmed breast abscess and
* presenting at KK Women's and Children's Hospital, Singapore

Exclusion Criteria: Patients with:

* mastitis
* granulomatous mastitis
* breast fillers with infection
* ruptured abscess prior to intervention
* other interventions or bilateral breast infection

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast abscess in females
Study Population: females with breast abscess
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
recovery time | from diagnosis to date of documented recovery defined as resolution of abscess, assessed up to 2 years
  recovery time for the abscess to resolve

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore